CLINICAL TRIAL: NCT02582632
Title: An Open-Label, Single Arm Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir in Treatment-Naïve Adults With Genotype 1b Hepatitis C Virus (HCV) Without Cirrhosis (GARNET)
Brief Title: A Study to Evaluate Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir in Treatment-Naïve Hepatitis C Virus Genotype 1b-Infected Adults
Acronym: GARNET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-684; 2015-003370-33 (EudraCT Number)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Infection; Hepatitis C Virus
Keywords: Hepatitis C Virus; Interferon-Free; Ribavirin-Free; Hepatitis C; Hepatitis C Genotype 1b
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; paritaprevir; dasabuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir (Experimental): Ombitasvir/Paritaprevir/Ritonavir(25 mg/150 mg/100 mg once daily) and Dasabuvir (250 mg twice daily) administered for 8 weeks
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: dasabuvir

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir — Tablet
  Other Names: ABT-267/ABT-450/r; ombitasvir also known as ABT-267; paritaprevir also known as ABT-450
Drug: dasabuvir — Tablet
  Other Names: ABT-333

SUMMARY:
This study will evaluate the safety and efficacy of ombitasvir/paritaprevir/ ritonavir and dasabuvir administered for 8 weeks in treatment-naïve participants with genotype 1b (GT1b) hepatitis C virus (HCV).

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HCV infection at Screening.
2. Screening laboratory result indicating HCV genotype 1b infection.
3. Treatment-naïve and non-cirrhotic.

Exclusion Criteria:

1. HCV genotype or subtype other than GT1b.
2. Positive test result for Hepatitis B surface antigen (HbsAg) or confirmed positive anti-HIV antibody (HIV Ab) test.
3. Any current or past clinical evidence of cirrhosis.
4. Screening laboratory analyses that shows abnormal results.
5. Clinically significant abnormalities or co-morbidities, other than HCV infection that make the participant an unsuitable candidate for this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-11-24; Primary Completion 2016-08-24 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dumas, PhD, Study Director — AbbVie

REFERENCES:
- [Background] Welzel TM, Asselah T, Dumas EO, Zeuzem S, Shaw D, Hazzan R, Forns X, Pilot-Matias T, Lu W, Cohen DE, Feld JJ. Ombitasvir, paritaprevir, and ritonavir plus dasabuvir for 8 weeks in previously untreated patients with hepatitis C virus genotype 1b infection without cirrhosis (GARNET): a single-arm, open-label, phase 3b trial. Lancet Gastroenterol Hepatol. 2017 Jul;2(7):494-500. doi: 10.1016/S2468-1253(17)30071-7. Epub 2017 Apr 14. PMID 28416221

RESULTS

PARTICIPANT FLOW:
Groups:
- Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir: ombitasvir/paritaprevir/ritonavir (25 mg/150 mg/100 mg once daily) and dasabuvir (250 mg twice daily) administered for 8 weeks
Period: Overall Study
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Started | 166
Completed | 165
Not Completed | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantification (LLOQ) 12 weeks after the last dose of study drugs without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. Confidence interval calculated using the normal approximation to the binomial distribution.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent to Treat (ITT) population: all enrolled participants who received at least 1 dose of study drug. Flanking imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 166
percentage of participants | 97.6 [95.3 to 99.9]

2. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Failure During Treatment Period
Description: On-treatment virologic failure is defined as breakthrough (confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment, or confirmed increase from nadir in HCV RNA (two consecutive HCV rna measurements > 1 log^10 IU/mL above nadir) at any time point during treatment) or failure to suppress during treatment (all on-treatment values of HCV RNA ≥ LLOQ) with at least 6 weeks (defined as study drug duration ≥ 36 days) of treatment. Confidence interval calculated using the normal approximation to the binomial distribution.
Time Frame: Up to 8 weeks while on treatment
Population: ITT population: all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 166
percentage of participants | 0.6 [0.0 to 1.8]

3. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse12
Description: Relapse12 is defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of active study drug (up to and including the SVR12 window) excluding reinfection among participants with HCV RNA < LLOQ at final treatment visit who complete treatment and have post-treatment HCV RNA data. Completion of treatment is defined as a study drug duration ≥ 51 days for participants who receive 8 weeks of treatment. HCV reinfection is defined as confirmed HCV RNA ≥ LLOQ after the end of treatment in a participant who had HCV RNA < LLOQ at final treatment visit, along with the post treatment detection of a different HCV genotype, subtype, or clade compared with baseline, as determined by phylogenetic analysis of the NS3 or NS5A, and/or NS5B gene sequences. Confidence interval calculated using the normal approximation to the binomial distribution.
Time Frame: Up to 12 weeks after last dose of study drug
Population: ITT population: all enrolled participants who received at least 1 dose of study drug. Participants who did not complete treatment or had no post treatment data available or had HCV RNA ≥ LLOQ at the Final Treatment Visit were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 163
percentage of participants | 1.2 [0.0 to 2.9]

4. Secondary Outcome: Percentage of Female Participants Responding With SVR12
Description: SVR12 is defined as HCV RNA < LLOQ 12 weeks after the last dose of study drugs without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. Confidence interval calculated using the normal approximation to the binomial distribution.
Time Frame: 12 weeks after the last actual dose of study drug
Population: ITT population: all enrolled female participants who received at least 1 dose of study drug. Flanking imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 94
percentage of participants | 97.9 [95.0 to 100.0]

5. Secondary Outcome: Percentage of Participants With Baseline HCV RNA < 6,000,000 IU/mL Responding With SVR12
Description: as for outcome 4
Time Frame: Baseline and 12 weeks after the last actual dose of study drug
Population: ITT population: all enrolled participants who received at least 1 dose of study drug and with baseline HCV RNA < 6,000,000 IU/mL. Flanking imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 154
percentage of participants | 98.1 [95.9 to 100.0]

6. Other Pre Specified Outcome: Percentage of Participants Who Achieve SVR12: mITT-GT Population
Description: as for outcome 4
Time Frame: 12 weeks after the last actual dose of study drug
Population: The modified ITT (mITT)-GT population includes participants who received at least 1 dose of study drug but excludes the participants who do not have HCV GT1b infection. Flanking imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 163
percentage of participants | 98.2 [96.1 to 100.0]

7. Other Pre Specified Outcome: Percentage of Participants With On-Treatment Virologic Failure During Treatment Period: mITT-GT Population
Description: On-treatment virologic failure is defined as breakthrough (confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment, or confirmed increase from nadir in HCV RNA (two consecutive HCV rna measurements > 1 log^10 IU/mL above nadir) at any time point during treatment) or failure to suppress during treatment (all on-treatment values of HCV RNA ≥ LLOQ) with at least 6 weeks (defined as study drug duration ≥ 36 days) of treatment. Confidence interval calculated using the Wilson score method.
Time Frame: Up to 8 weeks while on treatment
Population: The mITT-GT population includes participants who received at least 1 dose of study drug but excludes the participants who do not have HCV GT1b infection.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 163
percentage of participants | 0 [0.0 to 2.3]

8. Other Pre Specified Outcome: Percentage of Participants With Post-Treatment Relapse12: mITT-GT Population
Description: as for outcome 3
Time Frame: Up to 12 weeks after last dose of study drug
Population: The mITT-GT population includes participants who received at least 1 dose of study drug but excludes the participants who do not have HCV GT1b infection. Participants who did not complete treatment or had no post treatment data available or had HCV RNA ≥ LLOQ at the Final Treatment Visit were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 161
percentage of participants | 1.2 [0.0 to 3.0]

9. Other Pre Specified Outcome: Percentage of Female Participants Responding With SVR12: mITT-GT Population
Description: as for outcome 4
Time Frame: 12 weeks after the last actual dose of study drug
Population: The mITT-GT population includes participants who received at least 1 dose of study drug but excludes the participants who do not have HCV GT1b infection; female participants. Flanking imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 93
percentage of participants | 97.8 [94.9 to 100.0]

10. Other Pre Specified Outcome: Percentage of Participants With Baseline HCV RNA < 6,000,000 IU/mL Responding With SVR12: mITT-GT Population
Description: as for outcome 4
Time Frame: Baseline and 12 weeks after the last actual dose of study drug
Population: The mITT-GT population includes participants who received at least 1 dose of study drug but excludes the participants who do not have HCV GT1b infection; participants with baseline HCV RNA < 6,000,000 IU/mL. Flanking imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Number analyzed (Participants) | 151
percentage of participants | 98.7 [96.9 to 100.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 12 weeks); serious adverse events (SAEs) were collected from the time informed consent was obtained (up to 35 days prior to first dose of study drug).
Description: A TEAE is defined as any adverse event from the first dose of study drug to 30 days after the last dose.
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Serious Adverse Events (participants affected / at risk) | 2/166
Other Adverse Events (participants affected / at risk) | 70/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir (N=166)
GASTROENTERITIS (Infections and infestations) | 1
SYNCOPE (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir (N=166)
NAUSEA (Gastrointestinal disorders) | 11
ASTHENIA (General disorders) | 9
FATIGUE (General disorders) | 28
NASOPHARYNGITIS (Infections and infestations) | 14
HEADACHE (Nervous system disorders) | 35
PRURITUS (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.